CLINICAL TRIAL: NCT05276115
Title: An Experiential, One-to-one Interview Process Examining the Perception of Research Assessments and Equipment From Individuals With Post-traumatic Stress Disorder (PTSD)
Brief Title: PTSD Interview Regarding Future Study Design and Equipment.
Status: Suspended | Type: Observational
Why Stopped: Prioritizing other studies
Sponsor: Life University (Other)
Responsible Party: Sponsor
Other Study IDs: I-0018
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Ptsd
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Interview discussion with individuals with ptsd.

SUMMARY:
To gain insight and perspective unique to individuals with a diagnosis of PTSD, this study will utilize an experiential one-to-one interview format. During the interview, an investigator will walk the participants through several aspects of an ANS battery of tests, provide a tour and information about other equipment in the research lab and discuss tools and procedures associated with the application of chiropractic care. The aim of this research is to provide insight for future study designs that assess or provide care to individuals with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as having been diagnosed with PTSD.
* Between the ages 21-65 years old.

Exclusion Criteria:

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be included if they meet the following criteria:
  * Self-identify as having been diagnosed with PTSD.
  * Between the ages 21-65 years old.
  * Total of 15 individuals
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-11-17 (Estimated); Study Completion 2023-11-17 (Estimated)

PRIMARY OUTCOMES:
Interview | 1-2 hours
  Notes and further insights regarding individuals with PTSD's feelings toward the research space and the research equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Atlanta, Georgia, United States